CLINICAL TRIAL: NCT06263634
Title: Investigation of the Effect of Hand Exercises on Grip Strength, Functionality, Disease Activity and Quality of Life in Patients With Psoriatic Arthritis
Brief Title: Hand Exercises in Psoriatic Arthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Akdeniz University (Other)
Responsible Party: Principal Investigator, Sebahat Yaprak Cetin, PT, Principal Investigator, Akdeniz University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022-206
Record Dates: First submitted 2024-02-09; First posted 2024-02-16 (Actual); Last update posted 2024-06-10 (Actual); Status verified 2024-02

CONDITIONS: Psoriatic Arthritis; Hand Rheumatism
Keywords: Psoriatic Arthritis; hand exercises; grip strength; functionality; disease activity; quality of life
MeSH Terms: conditions — Arthritis, Psoriatic

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Home exercises group (Experimental): The intervention group will perform 30-45 minutes of home exercises consisting of stretching, mobility and strengthening, 4 days a week for 8 weeks, and the patients' compliance with the exercise will be monitored by phone call once a week.
  Interventions: Other: Hand exercises
- Control group (No Intervention): Patients in the control group will be on the waiting list and will be taught hand exercises when the program ends.

INTERVENTIONS:
Other: Hand exercises — 30-45 minutes of home exercises consisting of stretching, mobility and strengthening
  Arms: Home exercises group

SUMMARY:
This study is a randomized controlled study examining the effects of 8-week hand home exercises on grip strength, functionality, disease activity and quality of life in patients with PsA. Individuals participating in the study will be randomly divided into 2 groups. Individuals in the intervention group will perform home exercises consisting of stretching, mobility and strengthening, 4 days a week for 8 weeks, and the patients' compliance with the exercise will be monitored by phone call once a week. Individuals in the control group are on the waiting list and the same home exercise program will be taught to the patients at the end of the study.

DETAILED DESCRIPTION:
Psoriatic arthritis (PsA) is a chronic inflammatory musculoskeletal disease that is in the spondyloarthritis group and is frequently accompanied by peripheral arthritis, dactylitis, enthesitis, spondylitis and accompanied by psoriasis. Although hand effects in patients with PsA are known, there is no exercise study performed only on the hand and no study examining the effect of this study on the grip strength and functionality of the hand. This study is a randomized controlled study examining the effects of 8-week hand home exercises on grip strength, functionality, disease activity and quality of life in patients with PsA. 34 individuals with PsA who meet the inclusion criteria will be included in the study. Individuals participating in the study will be randomly divided into 2 groups. Individuals in the intervention group will perform 30-45 minutes of home exercises consisting of stretching, mobility and strengthening, 4 days a week for 8 weeks, and the patients' compliance with the exercise will be monitored by phone call once a week. Individuals in the control group are on the waiting list and the same home exercise program will be taught to the patients at the end of the study. Evaluations will be made twice, at the beginning and at the end of the 8-week program. In the evaluation, the demographic form, Psoriatic Arthritis Disease Activity Score (DAPSA), Grip Strength, Nine-Hole Peg Test, Duruöz Hand Index, Michigan Hand Outcome Questionnaire (MHQ) Functional Hand Index, Psoriatic Arthritis Quality of Life Questionnaire (PsAQoL) will be applied. This study will be one of the first studies to show the effects of hand exercises on PsA disease activity, grip strength, functionality and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Being diagnosed with PsA by a physician according to CASPAR criteria
* Being 18 years or older
* Involvement in hand joints (pain, swelling, tenderness)
* Being on stable drug treatment for the last 6 months
* Having sufficient cooperation to participate in the study
* Volunteering to participate in the study

Exclusion Criteria:

* Having difficulty cooperating at work
* Having additional orthopedic and/or neurological disease that will affect hand functions

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2023-04-05 (Actual); Primary Completion 2024-04-05 (Actual); Study Completion 2024-04-05 (Actual)

PRIMARY OUTCOMES:
Psoriatic Arthritis Disease Activity Score (DAPSA) | 8 weeks
  DAPSA; It is a composite measurement focused on peripheral arthritis, developed for reactive arthritis, adapted to PsA patients and frequently used, evaluating disease activity and response to treatment in clinical studies. There are four components of score including the parameters a) tender joint count (68 joints), b) swollen joint count (66 joints), c) CRP value (mg/l) and d) patient's disease activity and pain assessment (with a 10 cm visual analog scale). DAPSA scores are calculated by summing each of these components. Cut-off values for disease activity; A score of <4 was determined as remission, a score of <14 was determined as minimal disease activity, a score of <28 was determined as moderate disease activity, and a score of 28 was determined as high degree of disease activity.
Hand grip strength measurement | 8 weeks
  Hand grip strength will be measured with a Jamar hydraulic hand dynamometer (Sammons Preston, USA). Grip tests will be performed in the standard position recommended by the American Association of Hand Therapists. This is the standard position; The patient is seated in a position that provides 90-20 degree flexion of the hip and knee, shoulder adduction, forearm neutral position, 90 degree flexion of the elbow, 0-30 degree extension of the wrist and 0-15 degree ulnar deviation. The measurement will be repeated three times. There will be a 15-second rest break at the end of each measurement. As a result, the average of three measurements will be recorded.
Hand fine grip strength measurement: | 8 weeks
  Fine grip strength measurements will be made with finger dynamometry (Pinchmeter-Sammons Preston, USA). Grip tests will be performed in the standard position recommended by the American Association of Hand Therapists. This is the standard position; The patient is seated in a position that provides 90 degrees of hip and knee flexion, shoulder adduction, forearm neutral position, 90 degree flexion of the elbow, 0-30 degree extension of the wrist and 0-15 degree ulnar deviation. Three different finger grips will be evaluated. These:
  1- Fingertip grip strength, 2- Lateral grip strength, 3- Three point grip strength.
  Measurements will be repeated three times. There will be a 15-second rest break at the end of each measurement. As a result, the average of three measurements will be recorded.

SECONDARY OUTCOMES:
Nine-Hole Peg Test | 8 weeks
  This is a device consisting of a square platform and a storage box. There are 9 holes in the square-shaped area and 9 cylinders suitable for these holes. The patient is asked to quickly take the 9 cylinders from the storage box, place them in the holes in random order, and quickly remove them from the holes without taking a break and place them in the storage box. Meanwhile, time is measured in seconds with a stopwatch. The test is performed 2 times consecutively for both hands and the average of the result is taken. The total test score is calculated by averaging the scores for both hands.
Duruöz Hand Index | 8 weeks
  It is a valuable test that was first developed in 1996 to evaluate the hand functions of patients with Rheumatoid Arthritis and whose validity and reliability have been proven in many diseases related to the upper extremity. The test consists of 18 questions. It is a simple, useful and reliable test that is presented by separating daily life functions (kitchen, clothing, cleaning, workplace and other daily life activities), does not require additional training and equipment for the test, and takes approximately 2-3 minutes to apply. It is a simple and understandable test in which questions are answered according to a Likert scale, with a minimum score of 0 and a maximum of 90 points. A lower score indicates a better functional state.
Michigan Hand Outcome Questionnaire (MHQ) | 8 weeks
  This questionnaire is a scale consisting of six sections and 57 different items. It helps us question how well patients perform tasks they frequently perform. The patient answers the questions according to the Likert measurement method, which gives values from one to five. While each section receives a score between zero and one hundred, zero represents the worst score and one hundred represents the best score in each section, except for pain. A higher score in the pain section indicates more pain. The first part measures the average function of the patient's right and left hands. The second part contains questions examining daily living activities for both hands. In the third section, activities performed with both hands are questioned. The fourth part aims to question pain for both hands. In the fifth part, both hands are questioned aesthetically, and in the sixth part, the extent to which both hands satisfy the patient is questioned.
Hand Functional Index (HFI) | 8 weeks
  The validity and reliability of the Hand Functional Index (the first 9 questions of the Keitel Functional Index) were conducted by Mehmet Tuncay Duruöz in 1998 in patients with Rheumatoid Arthritis. The test consists of 9 questions. Each question has a different score. The highest total score an individual can get in the test is 21 points, and the lowest total score is 2. As the total score decreases, the functionality of the individual's hand increases.
Psoriatic Arthritis Quality of Life Questionnaire (PsAQoL) | 8 weeks
  It is used to evaluate the effects of PsA on individuals' quality of life. If there is a change in PsAQoL scores after treatment, it means that the applied treatment has an impact on the quality of life. This scale consists of 20 questions and is a practical, easily and quickly applicable survey with yes/no answers. Scoring is made as "yes: 1", "no: 0". A high score indicates a low quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Sebahat Yaprak Cetin, PhD, Principal Investigator — Akdeniz University
Locations (1):
- Akdeniz University, Antalya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Plans, data and analysis will share with SPSS program with other researchers

REFERENCES:
- [Result] Candiri B, Talu B, Demirtas Karaoba D, Ozaltin GE, Yolbas S. Effect of psoriatic arthritis on the strength, proprioception, skill, coordination, and functional condition of the hand. Int J Rheum Dis. 2022 Jan;25(1):47-55. doi: 10.1111/1756-185X.14241. Epub 2021 Nov 24. PMID 34821039
- See also: full text — http://pubmed.ncbi.nlm.nih.gov/34821039/